CLINICAL TRIAL: NCT01919034
Title: Evaluating the Relationship of Morphine Consumption and Pain-related Molecules in Hepatic Surgical Patients
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Yen Chin Liu, Visiting Staff, Department of Anesthesiology Chief, National Cheng-Kung University Hospital
Other Study IDs: B-ER-102-026
Record Dates: First submitted 2013-07-26; First posted 2013-08-08 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Pain; Huntington Disease; Hepatic Surgery
Keywords: Interleukin-20, Thrombomodulin, Huntington disease, patient control analgesic
MeSH Terms: conditions — Pain; Huntington Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood will be sampling (15cc/time), iver tissue (10mm3)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients undergoing abdominal surgery: Patients undergoing abdominal surgery and using morphine pain control analgesia (PCA) device will be involved. Pre- and Post- operative (after anesthesia and at the end of surgery) blood sampling (total 30 ml) plus normal liver tissue (10mm3) e will be harvested. Above protein(TM, IL-20, HD) amount change will be measured (ELISA for TM, IL-20 (serum) or flowcytometry (white cells) for TM, HD, IL-20 expression, stain or blotting for skin tissue). Patients will be included in this branch to check the correlation between morphine consumption and protein expression. Pain questionnaire (BPI, McGill) will be applied for pain evaluation. 2-D gel analysis will also be applied to screen further possible molecules.

SUMMARY:
According to above basic findings, it is important to confirm those results in clinic. In this branch, the investigators will use patient control analgesic (PCA) device to investigate the consumption of morphine for patients undergoing hepatic surgery. Preoperative and postoperative (before and after surgery) blood will be sampling (15cc/time) and y liver tissue (10mm3) will be harvested to measure the expression of above molecules (TM, IL-20, HD). Pain questionnaire will also be applied to evaluate their pain control quality. Certainly, the morphine consumption and results from pain questionnaire will be correlated with the molecule amount to figure out possible relationship between morphine consumption and those molecules.

Patients undergoing abdominal surgery and using morphine pain control analgesia (PCA) device will be involved. Pre- and Post- operative (after anesthesia and at the end of surgery) blood sampling (total 30 ml) plus normal liver tissue (10mm3) e will be harvested. Above protein(TM, IL-20, HD) amount change will be measured (ELISA for TM, IL-20 (serum) or flowcytometry (white cells) for TM, HD, IL-20 expression, stain or blotting for skin tissue). Patients will be included in this branch to check the correlation between morphine consumption and protein expression. Pain questionnaire (BPI, McGill) will be applied for pain evaluation. 2-D gel analysis will also be applied to screen further possible molecules.

Specific aims

1. To investigate the correlation of morphine consumption and the serum amount of IL-20, TM or HD
2. To investigate the relationship between IL-20, TM, HD amount in liver tissue and morphine consumption

DETAILED DESCRIPTION:
As the investigators all know, pain, as an ancient enemy to human kind, was one of the most mystical phenomena within our body. For centuries, people search the magic wand to solve this issue and reach the heaven destination. However, like our original sin commit by Adam and Eve, the shadow of pain always surround and even rebel our body and spirit. Even more, pain traps our soul and body not only for the acute stage induced by noxious stimulation but also change our mind and body whenever chronic period start even the stimulation disappears. Pain so far has become one of the greatest health issues for modern people. It affects millions of people and the treatment options are quite limited and not effective everyone. Drugs for pain relief are quite few kinds and associated with lots of side effect. On the other way, why and how people develop chronic pain, especially when there is no further painful stimulation, remain to be investigated. The integrated project, combining with our preliminary study and novel findings in our university (TM, IL-20, HD), will not only set a platform for pain drug discovery and their possible pathway in pain mechanism but also provide important clinical data for patients with severe pain under major surgery. Four sub-projects were included in this integrated project: 1. IL-20 is important in analgesia and pain mechanism. 2. the potential of thrombomodulin as an analgesic. 3. Huntington mice produce less pain behavior. 4. The relationship of morphine consumption and TM, IL-20 and HD protein for post-operative patients.

1.Interleukin-20 (IL-20) is a proinflammatory cytokine belonging to the IL-10 family. IL-20 is produced by activated keratinocytes and monocytes and transmits an intracellular signal through two distinct cell-surface receptor complexes on keratinocytes and other epithelial cells. IL-20 regulates proliferation and differentiation of keratinocytes during inflammation, particularly inflammation associated with the skin. It is also involved in the pathogenesis of osteoporosis and is a new target to treat this disease. However, little data demonstrated its role on pain. Meanwhile, IL-10 was involved many pain models and suppresses IL-10 expression also reduce pain in animal models. In this sub-project, Our preliminary data demonstrated increase of IL-20 after morphine administration. Therefore, the investigators will explore the role of IL-20 in pain management.

2.)Thrombomodulin(TM) is a transmembranous glycoprotein, thrombin mediating formation of active protein C (APC) which involving proinflammatory and procoagulant process. Thrombomodulin- thrombin complex activate protein C and inhibits coagulation cascade. Lectin-like domain (D1) of TM prevents neutrophil and monocyte adhesion with inhibiting inflammation process. In addition, TM bind with HMGB1 (high-mobility group box 1) and prevent leukocyte activation demonstrated in previous study. HMGB1 appears to have a role in neuropathic pain involving dorsal root ganglion and peripheral nerve injury in recent investigations and develop many therapies aim to HMGB1 including antibody in recent days. HMGB1 interact with RAGE and related to induce hyperalgesia in a rodent model of neuropathic pain and pain hypersensitivity after peripheral nerve injury. In this branch study, the investigators will use various pain models to evaluate the expression of TM in tissues.

3.Huntington disease(HD) is neurodegenerative genetic disorder that affects muscle coordination. It caused by autosomal dominant mutation in Huntingtin gene and accumulates Huntington protein. This protein plays an important role in nerve cells. It upregulates Brain Derived Neurotrophic Factor (BDNF) and essential for development. It is associated with vesicles and microtubules and involved in vesicle trafficking. It also interact with over 100 other protein. However, less investigation focuses this protein on pain sensory level. Under the cooperation of Dr. Yang, the investigators will investigate the over-expression Huntington protein mice that will induce Huntington disease. The investigators will work on this issue and deepen our finding and produce a new view for this old disease.

4.According to above basic findings, it is important to confirm those results in clinic. In this branch, the investigators will use the patient control analgesic (PCA) device to investigate the consumption of morphine for patients undergoing hepatic surgery. Preoperative and postoperative blood will be sampling and tinny liver tissue (10mm3) will be harvested to correlate their morphine consumption and pain questionnaire will be evaluated for their pain control quality. Certainly, the morphine consumption will be correlated with the molecule amount to figure out possible relationship between morphine consumption and those molecules.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with resectable liver tumor and are over 18 years of age.
2. Patients who present the will for his/her liver resection.
3. Patients who are competent to understand the study and provide written informed consent and participate in outcome measurements.

Exclusion Criteria:

* Patients have previous liver surgery. Patients are over 65 years of age. Patients are unable to read or write the pain questionaire, any condition that could interfere with the interpretation of outcome assessments, pregnant or lactating women or allergy to morphine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing liver surgery and using morphine pain control analgesia (PCA) device will be involved.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
consumption of morphine for patients undergoing hepatic surgery | 20 months
  Preoperative and postoperative blood will be sampling and tinny liver tissue (10mm3) will be harvested to correlate their morphine consumption will be evaluated for their pain control quality.

SECONDARY OUTCOMES:
various pain models of TM in tissues | 20 months
  The investigators will use various pain models to evaluate the expression of TM in tissues. Pre- and Post- operative (after anesthesia and at the end of surgery) blood sampling (total 30 ml) plus normal liver tissue (10mm3) e will be harvested. Above protein(TM, IL-20, HD) amount change will be measured (ELISA for TM, IL-20 (serum) or flowcytometry (white cells) for TM, HD, IL-20 expression, stain or blotting for skin tissue).
HD over-expressed mice and pain behavior | 20 months
  The investigators will work on HD over-expressed mice and pain behavior with morphine.
Change of IL-20 after morphine administration | 20 months
  Interleukin-20 (IL-20) is a proinflammatory cytokine belonging to the IL-10 family. IL-20 is produced by activated keratinocytes and monocytes and transmits an intracellular signal through two distinct cell-surface receptor complexes on keratinocytes and other epithelial cells. IL-20 regulates proliferation and differentiation of keratinocytes during inflammation, particularly inflammation associated with the skin. It is also involved in the pathogenesis of osteoporosis and is a new target to treat this disease.

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Chin Liu, Doctor, Study Chair — Department of Anesthesiology, National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Shengli Rd, Taiwan